CLINICAL TRIAL: NCT05489705
Title: Deliver Insights in Hypertrophic Cardiomyopathy and Observational Outcomes in Real World: United States and European Prospective Registry Study
Brief Title: A Prospective Registry Study to Assess Real-world Patient Characteristics, Treatment Patterns, and Longitudinal Outcomes in Patients Receiving Mavacamten and Other Treatments for Symptomatic Obstructive Hypertrophic Cardiomyopathy (Obstructive-HCM)
Acronym: DISCOVER-HCM
Status: Recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV027-012
Record Dates: First submitted 2022-08-03; First posted 2022-08-05 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Obstructive Hypertrophic Cardiomyopathy
Keywords: Obstructive hypertrophic cardiomyopathy; Obstructive HCM (oHCM); Mavacamten; Heart failure; oHCM
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Heart Failure | interventions — MYK-461

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mavacamten: Participants will receive mavacamten as prescribed by a physician according to standard of care for symptomatic oHCM
  Interventions: Drug: Mavacamten
- Beta-blocker (BB) / non-dihydropyridine (non-DHP) calcium channel blocker (CCB) / disopyramide: Participants will receive BB/non-DHP CCB/disopyramide as prescribed by a physician according to standard of care for symptomatic oHCM
  Interventions: Drug: Non-mavacamten symptomatic oHCM therapy

INTERVENTIONS:
Drug: Mavacamten — As per product label
  Groups: Mavacamten
Drug: Non-mavacamten symptomatic oHCM therapy — Including Beta-blocker (BB), non-dihydropyridine (non-DHP) calcium channel blocker (CCB) and/or disopyramide as per product label
  Groups: Beta-blocker (BB) / non-dihydropyridine (non-DHP) calcium channel blocker (CCB) / disopyramide

SUMMARY:
This registry evaluates patient characteristics, real-world treatment patterns, and short- and long-term outcomes in a population of patients in the United States and Europe with symptomatic obstructive hypertrophic cardiomyopathy (HCM) who are receiving mavacamten, receiving other treatment for obstructive HCM, or not receiving treatment for obstructive HCM due to intolerance or failure of prior treatment.

United States Sub-Study: The purpose of this study is to evaluate the safety of mavacamten in patients with symptomatic obstructive HCM in the real-world setting.

Europe Sub-Study: The purpose of this study is to evaluate the effectiveness and safety of mavacamten in patients with symptomatic obstructive HCM in the real-world setting.

ELIGIBILITY:
Inclusion Criteria

* ≥ 18 years of age at the time of informed consent.
* Willing and able to provide written informed consent form (ICF) and any required privacy authorization prior to the initiation of study procedures (or in those situations where consent cannot be given by participants, consent provided by their legally acceptable representatives)

United States Sub-Study

* Diagnosis of obstructive HCM consistent with 2020 American Heart Association/American College of Cardiology (AHA/ACC) guidelines.

  * Obstructive HCM is defined clinically by the presence of increased LV wall thickness ≥ 15 mm (or ≥ 13 mm with positive family history of HCM) in a nondilated ventricular chamber that is not solely explained by abnormal loading conditions (eg, another cardiac or systemic disease) and peak LVOT gradient of ≥ 30 mmHg at rest or with provocation.
* Has documented LVEF of ≥ 55% recorded by echocardiography within the last 6 months.
* Symptoms consistent with NYHA functional class II-IV.
* Receiving beta blocker (BB)s, non-dihydropyridine calcium. channel blockers (nonDHP CCBs), disopyramide, and/or mavacamten (once available) as part of routine clinical care; or currently receiving no treatment due to intolerance or failure of prior treatment (eg, BBs, non-DHP CCBs, or disopyramide) for obstructive HCM.

European Sub-study

* Diagnosis of obstructive HCM consistent with the most recent European Society of Cardiology (ESC) and American Heart Association/American College of Cardiology (AHA/ACC) guidelines
* Documented LVEF of ≥55% recorded by TTE
* Documented symptoms consistent with NYHA functional class II-III at enrollment or within 6 months prior to enrollment (if not available at enrollment).
* As part of routine clinical care for obstructive HCM: receiving BBs, non-DHP CCBs, disopyramide; initiating mavacamten at enrollment; or currently receiving no treatment due to intolerance or failure of prior treatment (e.g., BBs, non-DHP CCBs, or disopyramide).

Exclusion Criteria

* Known phenocopy disease (e.g., Fabry disease, amyloidosis) or LV hypertrophy associated with hypertension.
* Documentation of any fixed obstruction of the outflow tract such as aortic valve stenosis or replacement.
* Prior treatment of obstructive HCM with invasive septal reduction (surgical myectomy or percutaneous alcohol septal ablation [ASA]) within 6 months prior to enrollment; participants with an unsuccessful myectomy or percutaneous ASA performed > 6 months prior to enrollment may be enrolled.
* Naïve to treatment for obstructive HCM (ie, never treated with BBs, nonDHP CCBs, or disopyramide).

United States Sub-Study

* Receiving an investigational therapeutic agent for obstructive HCM (eg, myosin-inhibitors other than mavacamten) in an interventional clinical trial at participant enrollment.
* Previously or currently enrolled in a long-term safety extension study of mavacamten (eg, EXPLORER-HCM [ClinicalTrials.gov, NCT03470545], MAVA-LTE [NCT03723655], PIONEER-OLE [NCT03496168], VALORHCM [NCT04349072], or MAVERICK [NCT03442764])

European Sub-study

* Receiving an investigational therapeutic agent or any cardiac myosin inhibitor and/or modulators for obstructive HCM at patient enrolment
* Previously or currently enrolled in other HCM registry studies (e.g., TORCH, REMY, EU-PASS)
* Previously or currently enrolled in a study of mavacamten (e.g., EXPLORER-HCM [ClinicalTrials.gov, NCT03470545], MAVA-LTE [NCT03723655], PIONEER-OLE [NCT03496168], VALOR-HCM [NCT04349072], MAVERICK [NCT03442764], or MEMENTO [NCT2264899])
* Previously treated with mavacamten

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adult participants with symptomatic obstructive HCM who are receiving pharmacological treatment for obstructive HCM (for example, BBs, non-DHP CCBs, disopyramide, and/or mavacamten) as part of routine care in the United States or Europe.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2022-08-16 (Actual); Primary Completion 2029-08-17 (Estimated); Study Completion 2029-08-17 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of new or worsening heart failure due to systolic dysfunction among participants with symptomatic obstructive HCM during periods of exposure to mavacamten and other oHCM treatment | Up to 5 Years
  Systolic dysfunction defined as symptomatic Left Ventricular Ejection Fraction (LVEF) < 50%. United States participants only.
Change in resting left ventricular outflow tract (LVOT) gradient from baseline | Up to 18 months
  European Participants only

SECONDARY OUTCOMES:
Occurrence of arrhythmia | Baseline, and up to 18 months (European participants), or 5 Years (United States participants)
  Incidence rates of participants with arrhythmia (new onset)
New or worsening heart failure due to systolic dysfunction | Baseline and up to 18 months
  Symptomatic left ventricular ejection fraction (LVEF) <50%. European Participants only
Proportion of participants with a resting or provoked peak left ventricular outflow tract (LVOT) gradient below 50 mmHG | Baseline and up to 18 months
  European participants only
Proportion of participants with a resting or provoked peak left ventricular outflow tract (LVOT) gradient below 30 mmHG | Baseline and up to 18 months
  European participants only
Occurrence of Major Adverse Cardiovascular Events (MACE) | Up to 5 Years
  A composite endpoint consisting of non-fatal acute Myocardial Infarction (MI), stroke, hospitalization due to Heart Failure (HF) and Cardiovascular (CV) mortality. United States participants only.
Occurrence of non-fatal acute Myocardial Infarction (MI) | Up to 5 Years
  United States participants only
Occurrence of Stroke | Up to 5 Years
  United States participants only
Occurrence of hospitalization due to heart failure | Baseline, and up to 18 months (European participants), or 5 Years (United States participants)
Occurrence of cardiovascular mortality | Up to 5 Years
  United States participants only
Occurrence of all-cause mortality | Baseline, and up to 18 months (European participants), or 5 Years (United States participants)
Evaluation of functional responses: New York Heart Association (NYHA) function class | Baseline, and up to 18 months (European participants), or 5 Years (United States participants)
  Percentage of Participants Whose NYHA Class Changes
Evaluation of functional responses: Left Ventricular Outflow Tract (LVOT) gradient | Baseline, and up to 18 months (European participants), or 5 Years (United States participants)
  Mean Change From Baseline in LVOT Gradients At Rest and Provoked
Evaluation of functional responses: LVEF | Baseline, and up to 18 months (European participants), or 5 Years (United States participants)
  Mean Change from Baseline in LVEF
Evaluation of patient reported outcome measure: Kansas City Cardiomyopathy Questionnaire 23 (KCCQ-23) | Baseline, and up to 5 Years
  The KCCQ-23 is a disease-specific health status instrument composed of 23 items that quantifies the domains of physical limitations, symptoms, self-efficacy, social limitation and quality of life from heart failure. Scores range from 0-100, in which higher scores reflect better health status. United States participants only
Evaluation of patient reported outcome measure: EuroQol Five Dimensions Questionnaire (5-level) (EQ-5D-5L): Health Utility Index | Baseline, and up to 5 Years
  The EQ-5D-5L is a 2-part instrument for use as a measure of health outcome, designed for self-completion by respondents. It consists of EQ-5D-5L health utility index and EQ Visual Analog Scale (VAS). EQ-5D-5L health utility index is comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each has 5 levels of perceived problems (1-no problem, 2-slight problems, 3-moderate problems, 4-severe problems, 5-extreme problems). Participants select an answer for each of the 5 dimensions that best matches his/her health "today". Responses are used to generate a weighted summary index, which ranges from 0 to 1.00. A higher score indicates better health and positive changes from baseline indicate improvement of health. United States participants only
Evaluation of patient reported outcome measure: EQ-5D-5L: VAS | Baseline, and up to 5 Years
  The EQ-5D-5L is a 2-part instrument for use as a measure of health outcome, designed for self-completion by respondents. It consists of EQ-5D-5L descriptive system and VAS.
  The VAS self-rating records the participant's own assessment of his or her overall health status at the time of completion, on a vertical line VAS with scale of 0 (the worst health you can imagine) to 100 (the best health you can imagine). A higher score indicates better health and positive changes from baseline indicate improvement of health status. United States participants only
Evaluation of biomarkers of response: NT-proBNP | Baseline, and up to 5 Years
  Change From Baseline in Serum concentration of NT-proBNP. United States participants only
Evaluation of biomarkers of response: Cardiac troponin | Baseline, and up to 5 Years
  Change From Baseline in Serum Concentration of Cardiac Troponins. United States participants only

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (99):
- United States (62):
  - Alaska Heart Institute, Anchorage, Alaska
  - Pima Heart and Vascular, Tucson, Arizona
  - UAMS, Little Rock, Arkansas
  - UC San Diego School of Medicine, La Jolla, California
  - Keck School of Medicine of USC-Usc, Los Angeles, California
  - Stanford Health Care Hospital & Clinics, Palo Alto, California
  - University Of California San Francisco Medical Center, San Francisco, California
  - UC Denver, AMC, Aurora, Colorado
  - Hartford HealthCare, Hartford, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Uf Health Jacksonville, Jacksonville, Florida
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - University of Chicago Dept of Medicine, Chicago, Illinois
  - Indiana. University, Indianapolis, Indiana
  - Franciscan Physician Network-Indiana Heart Physicians, Indianapolis, Indiana
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - University Of Kansas Medical Center & Medical Pavilion, Kansas City, Kansas
  - University Of Maryland, Ihv, Baltimore, Maryland
  - MedStar Health Research Institute, Baltimore, Maryland
  - Harvard (Massachusetts General Hospital), Boston, Massachusetts
  - Harvard Medical School - Brigham and Women's Hospital (BWH), Boston, Massachusetts
  - Spectrum Health Medical Group, Grand Rapids, Michigan
  - Henry Ford Health System, West Bloomfield, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Cardiology Associates Research, Llc, Tupelo, Mississippi
  - St. Luke's Mid-America Heart Institute, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - CHI Health Reseach Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Bassett Medical Center, Cooperstown, New York
  - Northwell Health, Manhasset, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Saint Francis Hospital, Roslyn, New York
  - WMCHealth Advanced Physician Services, Valhalla, New York
  - Focus Clinical Research, Charlotte, North Carolina
  - Duke University Health System, Durham, North Carolina
  - Christ Hospital Health Network, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - AHN Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University Of Pittsburgh, Pittsburgh, Pennsylvania
  - Geisinger Health System, Wilkes-Barre, Pennsylvania
  - Prisma Health - Upstate, Greenville, South Carolina
  - Tristar Centennial Medical Ctr, Nashville, Tennessee
  - Saint Thomas Health, Nashville, Tennessee
  - North Texas Cardiology Center, Dallas, Texas
  - Baylor Scott & White Research Institute, Dallas, Texas
  - The Methodist Hospital, Methodist Cancer Cencer, Houston, Texas
  - BI Research Center, Houston, Texas
  - Baylor Scott & White The Heart Hospital Plano, Plano, Texas
  - Baylor Scott & White Medical Centre - Temple, Temple, Texas
  - The Rector and Visitors of the Univ of Virginia, Charlottesville, Virginia
  - VCU Medical Center, Richmond, Virginia
  - Carilion Clinic; Virginia Tech-Carilion School of Medicine, Roanoke, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - WVU Hospitals, Morgantown, West Virginia
  - University Of Wisconsin - Madison, Madison, Wisconsin
  - Medical College of Wisconsin, Inc (PI Address), Milwaukee, Wisconsin
- Austria (7):
  - KH St.Josef Braunau am Inn, Braunau am Inn
  - LKH-Univ. Klinikum Graz, Graz
  - Local Institution - 0088, Innsbruck
  - Local Institution - 0084, Klagenfurt
  - Kepler Universitätsklinikum Linz, Linz
  - Local Institution - 0085, Sankt Pölten
  - Local Institution - 0083, Vienna
- France (7):
  - Centre Hospitalier Haguenau, Haguenau, Bas Rhin
  - CHU Nantes Hopital Nord Laennec, Saint-Herblain, Loire Atlantique
  - Hôpital Saint Vincent-de-Paul, Lille, Nord
  - CHU Amiens-Picardie, Amiens, Somme
  - Hôpital Sainte Musse, Toulon, Var
  - CHU De Poitiers - Hopital De La Miletrie, Poitiers, Vienne
  - Local Institution - 0117, Montpellier
- Germany (7):
  - Ostalb-Klinikum Aalen, Aalen, Baden-Wurttemberg
  - Local Institution - 0101, Erlangen, Bavaria
  - Universitatsklinikum Muenster, Münster, North Rhine-Westphalia
  - Praxisklinik Herz Und Gefasse-Klinikum Weisser Hirsch, Dresden, Saxony
  - Universitaetsklinikum Leipzig Aoer, Leipzig, Saxony
  - Immanuel Klinikum Bernau, Bernau, State of Berlin
  - Kardiologische und angiologische Praxen im Spreebogen, Berlin
- Research & Cardiovascular Corp, Ponce, Puerto Rico
- Spain (8):
  - Hospital Fundacion Son Llatzer, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Virgen de La Arrixaca, El Palmar, Murcia
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario de Burgos, Burgos
  - Local Institution - 0102, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Clinico Universitario Virgen de La Victoria, Málaga
- United Kingdom (7):
  - Local Institution - 0113, London, Greater London
  - Imperial College Healthcare NHS Trust, London, Greater London
  - University Of Manchester, Manchester, Greater Manchester
  - Liverpool Heart and Chest Hospital, Liverpool, Merseyside
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham, West Midlands
  - Leeds General Infirmary, Leeds, West Yorkshire
  - University Hospital of Wales, Cardiff

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts